CLINICAL TRIAL: NCT03282409
Title: Prediction of Chronic Renal Disease After Acute Kidney Injury in the Intensive Care Unit
Acronym: PREDICT
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOR16089
Record Dates: First submitted 2017-07-31; First posted 2017-09-14 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Acute Kidney Injury; Chronic Renal Disease
Keywords: Prediction; Chronic Renal Disease; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to develop and validate a prediction score of chronic renal disease occurrence within 3 years after ICU discharge in patients who suffered an acute kidney failure during ICU stay and recovered normal renal function at 90 days following their discharge.

The primary study outcome is the incidence of chronic renal disease within the first 3 years after ICU discharge, defined by a lower glomerular filtration rate (GFR) under 60 mL/minute/1.73m2.

DETAILED DESCRIPTION:
As second objectives, the study aims to:

* Evaluate the GFR decline in patients who had an underlying chronic kidney disease.
* Evaluate factors associated with a persistent decreased GFR at day-90.
* Characterization the clinical and biological phenotype of chronic renal disease in these patients.
* Evaluate treatments provided to these patients according to CKD occurence.
* Evaluate the rate of cardiovascular and thrombo-embolic morbidity-mortality.
* Assess the quality of life every year for 3 years.
* Evaluate the medico-economic burden of CKD.

ELIGIBILITY:
Inclusion Criteria:

* Patient ⩾ 18 years;
* Patient suffering an acute kidney injury (defined by AKIN score ⩾1) during ICU stay;
* Patient discharged alive from the ICU;
* Patient's signed consent obtained;
* Patient covered by a healthcare insurance.

Exclusion Criteria:

* Pregnant or breastfeeding woman;
* SOFA score < 1 (except for kidney assessment) at time of ICU admission;
* End-stage of renal failure or dialysis treatment or renal transplantation prior to ICU admission;
* Patient treated with dialysis at ICU discharge;
* Immunosuppressive treatment prior to ICU admission;
* Patient under legal incapacity (tutor or guardian protection);
* Being unable to follow-up of the study;
* Life expectancy expected shorter than 90 days;
* Refusal to participate in the study;
* Patient's main address is outside of Il de France region for the centers in this region;
* Patient < 18 years;
* Patient not affiliated to national social security scheme;
* Patient deprived of liberty by judicial measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with acute kidney injury during ICU stay
Sampling Method: Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic kidney disease | At 3 years
  Incidence of chronic kidney disease defined by a decreased glomerular filtration rate (GFR) under 60 mL/minute/1.73m2.

SECONDARY OUTCOMES:
Progression of chronic renal disease defined by the slope of GFR decline | At 3 years
  For patients who have chronic renal disease history and developped an acute kidney failure during ICU stay, progression of chronic renal disease defined by a GFR decline greater than 30% at 3 years.
Progression of the proteinuria | At 3 years
  Evolution of urinary protein to creatinine ratio (mg/mmol).
Progression of chronic renal disease defined by the number of patients with end-stage renal disease requiring dialysis or renal transplantation | At 3 years
  For patients who have chronic renal disease history and developped an acute kidney failure during ICU stay, progression of chronic renal disease defined by need to dialysis, or need a renal transplantation, and GFR < 15mL/minute/1.73m2.
Occurrence of cardiovascular events and thromboembolic events | At 3 years
  Cardiovascular events include acute coronary syndrome, ischemic stroke, peripheral artery disease, ventricular rhythm disorder and sudden death.
  Thromboembolic events included deep vein thrombosis and pulmonary embolism.
All-cause mortality | At 3 years
  All-cause mortality and cardiovascular cause mortality
Quality of life assessment | At the end of 1 year
  Assessment of quality of life of patients by the scale KDQOL-SF-12. The SF-12 is a short form that includes Items 1-12 as generic core of kidney Disease Quality of Life Instrument (KDQOL).
Quality of life assessment | At the end of 1 year
  Assessment of quality of life of patients by the scale EQ-5D-5L. The EQ-5D-5L questionnaire consists the descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state.
Cost | At 3 years
  Costs related to medical care

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Geri, MD, PhD, Principal Investigator — Service de Réanimation médico-chirurgicale, Hôpital Ambroise Paré; Antoine Vieillard Baron, MD, PhD, Study Director — Service de Réanimation médico-chirurgicale, Hôpital Ambroise Paré
Locations (1):
- Intensive care unit, Ambroise Pare Hospital, Boulogne-Billancourt, Hauts-de-seine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Roquetaillade C, Durand M, Beaucote V, Guillemin J, Chadjichristos CE, Roquilly A, Chousterman BG. Progression of Kidney Fibrosis after Sepsis: Underestimated Role of Resident Macrophages and Recruited Monocytes. J Am Soc Nephrol. 2025 Mar 28;36(7):1417-1427. doi: 10.1681/ASN.0000000712. PMID 40152940
- [Derived] Geri G, Stengel B, Jacquelinet C, Aegerter P, Massy ZA, Vieillard-Baron A; PREDICT investigators. Prediction of chronic kidney disease after acute kidney injury in ICU patients: study protocol for the PREDICT multicenter prospective observational study. Ann Intensive Care. 2018 Jul 6;8(1):77. doi: 10.1186/s13613-018-0421-7. PMID 29980878